CLINICAL TRIAL: NCT02118844
Title: Laparoscopic Bariatric Surgery: Impact of the Level of Neuromuscular Blockade on Surgical Conditions - Comparison Between Moderate and Deep Neuromuscular Blockade
Brief Title: Laparoscopic Bariatric Surgery: Impact of Deep Neuromuscular Block on Surgical Conditions
Acronym: BaChiBloPro1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2014-000289-23
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Bariatric Surgery; Laparoscopic Bariatric Surgery; Robotic Bariatric Surgery; Gastric Bypass; Morbid Obesity
Keywords: bariatric surgery; surgical conditions; deep neuromuscular blockade
MeSH Terms: conditions — Obesity, Morbid | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderate rocuronium neuromuscular blockade (Active Comparator): rocuronium bolus is given if needed to maintain moderate neuromuscular blockade (TOF-count 2-4) during gastrojejunal anastomosis
  Interventions: Drug: rocuronium
- deep rocuronium neuromuscular blockade (Experimental): rocuronium bolus is given if needed to maintain deep neuromuscular blockade (here defined as a Posttetanic Count 1 - 5) during gastrojejunal anastomosis
  Interventions: Drug: rocuronium

INTERVENTIONS:
Drug: rocuronium

SUMMARY:
The purpose of this study is to determine whether deep neuromuscular blockade compared to moderate neuromuscular blockade may improve the surgical conditions in patients undergoing laparoscopic bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* patient between 18 and 64 years
* indication for bariatric surgery accordingly to HAS
* patient undergoing laparoscopic or robotic gastric bypass surgery
* written informed consent
* affiliation to social security

Non-inclusion Criteria:

* known hypersensibility to any of the drugs used during this study
* absence of written informed consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-08 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Improvement of surgical conditions | 15 minutes
  The surgical conditions will be evaluated with the King Score (M. King et al Anesthesiology 2000; 93: 1392 - 97). This score is a 4-point score. The evaluation will be done by the surgeon who is blinded. An improvement of at least 1-point will be considered as clinical relevant.

SECONDARY OUTCOMES:
Pneumoperitoneum generated pressure | 15 minutes
  Concomitantly to the evaluation of the surgical conditions the pneumoperitoneal pressure (in mm Hg) generated by the Carbon dioxide insufflation will be registrated.

OTHER OUTCOMES:
time needed to perform gastrojejunal anastomosis | 90 minutes
  The time from begin of the gastrojejunal anastomosis until the end will be measured in min. The surgeon indicate begin and end of the gastrojejunal anastomosis.
10 point-VAS to evaluate surgical conditions | 2 x 15 minutes
  Concomitantly the the evaluation by the King score, the surgical conditions will be also evaluated by a 10 point VAS (visual-analog scale).This evaluation will also be realized by the surgeon, still blinded to the study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Fuchs-Buder, MD, Principal Investigator — CHU Nancy, Department of Anaesthesia & Critical Care
Locations (1):
- CHU Nancy/Brabois, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Derived] Fuchs-Buder T, Schmartz D, Baumann C, Hilt L, Nomine-Criqui C, Meistelman C, Brunaud L. Deep neuromuscular blockade improves surgical conditions during gastric bypass surgery for morbid obesity: A randomised controlled trial. Eur J Anaesthesiol. 2019 Jul;36(7):486-493. doi: 10.1097/EJA.0000000000000996. PMID 30985536